CLINICAL TRIAL: NCT03061578
Title: A Clinical Study to Evaluate Innovative Tear Film Imaging for the Evaluation of Dry Eye and Its Correlation to Traditional Signs and Symptoms of Dry Eye Syndrome in a Low Humidity Environmental Exposure Chamber (LH-EEC)
Brief Title: Evaluation of Dry Eye by Tear Film Imager in a Low Humidity Environmental Exposure Chamber (TFI-LH16)
Acronym: TFI-LH16
Status: Completed | Type: Observational
Sponsor: Adom Advanced Optical Technologies Ltd. (Industry)
Collaborators: Inflamax Research Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: TFI-A2-LH-EEC-16
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Dry Eye
Keywords: Tear Film; Hyperspectral imaging; Low Humidity Environmental Exposure Chamber
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NDE: Non Dry Eye (NDE) group will be used as control for DES diagnosis.
  Subjects in the non-dry eye criteria must meet all of the following criteria:
  1. Have a Schirmer's Test (without anesthesia) of ≥10mm/5min in both eyes
  2. OSDI questionnaire score <13.
  3. Fluorescein TBUT > 7 s in both eyes.
  4. CFS of 0 in all areas in both eyes.
  The NDE group will undergo the same diagnosis including Tear Film Imager diagnostic and Low Humidity Environmental Exposure Chamber (LH-EEC) stimulation as any other group of patients.
  Interventions: Diagnostic Test: Tear Film Imager; Diagnostic Test: Low Humidity Environmental Exposure Chamber (LH-EEC)
- ADDE: Aqueous Deficiency Dry Eye (ADDE) group will be define by commonly known signs and symptoms.
  In order to classify subjects to the moderate to severe ADDE group, subjects must meet a predefined medical condition (Rheumatoid Arthritis, Dermatomyositis, Lupus or Sjögren's syndrome) and meet at least one of the following conditions:
  1. Have a Schirmer's Test (without anesthesia) of ≤5mm/5min in either eye
  2. Mean CFS of ≥1 in either eye.
  3. Fluorescein TBUT ≤5 s in either eye.
  4. OSDI questionnaire score ≥20
  The ADDE group will undergo the same diagnosis including Tear Film Imager diagnostic and Low Humidity Environmental Exposure Chamber (LH-EEC) stimulation as any other group of patients.
  Interventions: Diagnostic Test: Tear Film Imager; Diagnostic Test: Low Humidity Environmental Exposure Chamber (LH-EEC)
- LDDE: Lipid Deficiency Dry Eye (LDDE) group will be define by commonly known signs and symptoms.
  In order to classify subjects to the moderate to severe LDDE group, subjects must have moderate to severe Meibomian Gland Dysfunction (MGD score of 3-6) and meet at least one of the following conditions:
  1. Have a Schirmer's Test (without anesthesia) of ≤5mm/5min in either eye
  2. Mean CFS of ≥1 in either eye.
  3. Fluorescein TBUT ≤5 s in either eye.
  4. OSDI questionnaire score ≥20
  The LDDE group will undergo the same diagnosis including Tear Film Imager diagnostic and Low Humidity Environmental Exposure Chamber (LH-EEC) stimulation as any other group of patients.
  Interventions: Diagnostic Test: Tear Film Imager; Diagnostic Test: Low Humidity Environmental Exposure Chamber (LH-EEC)

INTERVENTIONS:
Diagnostic Test: Tear Film Imager — Ocular surface imaging assessment by the Tear Film Imager (TFI)
Diagnostic Test: Low Humidity Environmental Exposure Chamber (LH-EEC) — Subjects will enter the LH-EEC (<15% relative humidity (RH), temperature 22±5ºC, and 5±3ft/s directed air flow velocity) and remain for approximately 120 min.

SUMMARY:
The study consists of 3 study visits to the clinic over at least 9 days. Visit 1 - the medical screening visit: subjects will undergo informed consent and will be tested for signs and symptoms of Dry Eye Syndrome (DES) including measurements by the TFI.

Upon conclusion of the screening for DES, the subjects will be divided to the different categories: NDE, LDDE and ADDE. For ADDE and LDDE subjects the eye fitting the worst DES inclusion criteria will be designated as the study eye. For the NDE subjects the best eye will be designated as the study eye.

During Visit 2 and 3, the TFI measurement and other clinical study endpoint procedures will be only conducted on the study eye. The safety endpoint procedures will still be conducted on both eyes individually throughout the study. Subjects will be queried for adverse events (AEs) at all visits.

Visit 2 - after two days washout period subject will return for the LH-EEC test. Signs and symptoms of dry eye will be recorded before entering the LH-EEC, during the 120 min stay in the LH-EEC and at the conclusion of the day.

Visit 3 - after 7 days washout period subject will return for the last test. The third day procedure is identical to the second day, with the addition of: following LH-EEC exit, subjects will have a health check and study check out procedures conducted.

Statistical Analysis:

Data will be summarized with respect to baseline characteristics, efficacy variables and safety variables. Summary statistics will include the number of observations (N), mean, standard deviation (SD), median, minimum and maximum values for continuous variables and frequencies and percentages for categorical variables.

Missing values will not be replaced or imputed, i.e., no interpolation or extrapolation will be applied to missing values.

Safety data will be listed and summarized by group (NDE, ADDE, and LDDE).

DETAILED DESCRIPTION:
This study consists of 3 study visits to the clinic (a medical screening visit, and 2 LH-EEC visits) over at least 9 days. Subjects need to refrain from putting on any makeup near their eyes on the morning of each visit.

At the medical screening visit (Visit 1), subjects will undergo informed consent, fill out the Ocular Surface Disease Index (OSDI) questionnaire, and provide medical/surgical/ocular/medication histories and demographics. A urine pregnancy test will be performed on women of childbearing potential (WOCBP). Prior to any baseline symptom or sign collection, subjects will be acclimatized to the clinic environment for at least 30 min. Baseline subject rating of ocular symptoms (dryness, burning/stinging, tearing, grittiness/sandiness, intermittent blurring, soreness/discomfort, sensitivity to light [photophobia]) in both eyes together will be recorded using the electronic Patient Data Acquisition Tablet (ePDAT™) on a 0-4 scale with 0.5 increments. To meet eligibility criteria, subjects will participate in the following ophthalmic examinations (in the order specified): distance visual acuity (VA), slit lamp examination (SLE), undilated fundus examination, non-contact tonometry (NCT) followed by at least a 30 min wait, baseline TFI ocular surface imaging assessment (duplicate measurements at least 30 min apart in both eyes), Tear Break Up Time (TBUT), corneal fluorescein staining (CFS), conjunctival lissamine green staining (CLGS), Schirmer's Test without anesthetic, and Meibomian Gland Dysfunction (MGD)testing. Upon conclusion of the screening for DES, the eye fitting the worst DES inclusion criteria will be designated as the study eye. For the NDE subjects, the best eye will be designated as the study eye. During Visit 2 and 3, the TFI measurement and other clinical study endpoint procedures (i.e. TBUT, CFS, CLGS, Schirmer's Test) will be only conducted on the study eye, however the safety endpoint procedures (i.e. VA, SLE, undilated fundus exam NCT) will still be conducted on both eyes individually throughout the study. Subjects will be queried for adverse events (AEs) at all visits. The clinic environment will be monitored for relative humidity (%RH) and temperature (ºC) at each visit.

After at least a 2 day washout period, subjects will return to the clinic for Visit 2.

Prior to any baseline symptom or sign collection, subjects will be acclimatized to the clinic environment for at least 30 min. Subjects will be queried for changes in health and medication use since the last visit. Baseline subject rating of the 7 subjective ocular symptoms will be recorded using the ePDAT™. Baseline ophthalmic evaluations will be conducted (in the order specified) including VA, SLE followed by at least a 30 min wait, TFI assessment (single measurement only), TBUT, CFS, CLGS and Schirmer's Test without anesthetic. Following the Schirmer's Test, subjects will wait at least 60 min in the clinic and during this time, baseline blink rate (blink/min, in triplicate) will be measured. Subjects will then have a second TFI measurement and then enter the LH-EEC. Subject symptom scoring and staff assessed blink rate will be assessed on both eyes together throughout the study.

Subjects will enter the LH-EEC (<15% relative humidity (RH), temperature 22±5ºC, and 5±3ft/s directed air flow velocity) and remain for approximately 120 min. During this time subjects are asked to visually task on a digital screen to ensure the ocular surface is exposed to the airflow and humidity levels in the room. Environmental conditions in the LH-EEC, including relative humidity (%RH) and temperature (ºC), will be monitored. Subject-assessed symptoms will be assessed at 15, 30, 60, 90, and 120 min (+5 min), while in the LH-EEC. Blink rate and TFI tear film imaging assessment (single measurement on the study eye only) will be assessed by qualified staff at 35, 65, 95 min (+15 min), and prior to LH-EEC exit. After all other procedures and prior to exiting the chamber, VA, TBUT, CFS, CLGS, and Schirmer's Test without topical anesthetic, will be performed. After LH-EEC exit, a health check will be conducted.

After at least a 7 day washout period, subjects will return to the clinic on Visit 3 for their second LH-EEC visit. Subjects will be queried for changes in health and medication use since the last visit. Subjects will once again enter the LH-EEC (<15% relative humidity [RH], temperature 22±5ºC, and 5±3ft/s directed air flow velocity) for approximately 120 min. All procedures prior to LH-EEC entry, during LH-EEC exposure and prior to LH-EEC exit will be repeated as in Visit 2.

Following LH-EEC exit, subjects will have a health check and study check out procedures conducted including: VA, SLE, undilated fundus exam, and NCT.

Analysis Sets:

The Safety set will consist of all subjects who were enrolled in the study. The Modified Intent-to-Treat population (MITT) set will consist of all subjects who were enrolled in the study and who entered the LH-EEC and provided at least one post-baseline measurement. The Per-Protocol population (PP) set will consist of all subjects from MITT population who complete Visit 3 and do not have any protocol violations that may substantially affect the results.

Statistical Analysis:

Data will be summarized with respect to baseline characteristics, efficacy variables and safety variables. Summary statistics will include the number of observations (N), mean, standard deviation (SD), median, minimum and maximum values for continuous variables and frequencies and percentages for categorical variables. Missing values will not be replaced or imputed, i.e., no interpolation or extrapolation will be applied to missing values.

Safety data will be listed and summarized by group (NDE, ADDE, and LDDE). Any deviation(s) from the planned statistical analysis will be described and fully justified in the Statistical Analysis Plan (SAP) and/or the final clinical study report (CSR) as appropriate.

Demographic and Baseline Characteristics:

Demographic and baseline characteristics of subjects who participated in this study will be summarized by study group (NDE, ADDE, and LDDE) and overall using descriptive statistics. Distributions of these baseline parameters among study groups will be compared descriptively only. No statistical inference will be performed.

Safety Analysis:

Safety will be evaluated via the following parameters: AEs, SLE, VA, NCT, Fundus examination AEs will be summarized for severity and causality. AEs will be summarized by body system and preferred term within each study group (NDE/ADDE/LDDE). Each AE will be counted only once for a given subject. If the same AE occurred in a subject on multiple occasions, the highest severity and maximum causality relationship will be assumed. Serious AEs (SAEs), if any, will be summarized by body system, preferred term and study group. All AEs will be listed, along with SAEs and AEs leading to discontinuation. NCT assessment will be performed at Screening (Visit 1) and at end of study (Visit 3), to measure the Intra-Ocular Pressure (IOP). The collected data (average of 3 readings for each eye) will be listed by study group, subject and visit. Summary statistics of the average of 3 readings for each eye will be tabulated for Study eye, Right and Left eye. Study eye will be defined in the SAP. VA assessment will be performed at each visit. Data will be listed by ADDE/ LDDE/NDE group, subject and visit.

Statistical Study Termination:

If the device related SAE rate exceeds 20% in any specific group (ADDE/LDDE/NDE) the study of this group will be halted and a report will immediately be sent to the Sponsor. The Investigator and the Sponsor will analyze this report and offer a protocol update to the Institutional Review Board (IRB) to rectify the problem. If the IRB approves the updated protocol, the study will continue based on the updated protocol. If the IRB will not accept the updated protocol the specific group study will be terminated.

Analysis of the Endpoints:

The analyses of the clinical endpoints will be carried out using both the MITT and PP populations. All summary tables will be provided by study group (NDE, ADDE, and LDDE) and overall. The repeatability of the TFI will be evaluated from summary of TFI assessments between Visit 2 and Visit 3. The sensitivity of the imager to detect changes in ocular surface integrity will be evaluated from the summary of baseline to post baseline assessment scores by time points and visit. The correlation between the clinical measurements of DE and the corresponding TFI measurement of interest will evaluate the association between the two assessments. Descriptive statistics of all observed assessment scores at each time point and the change at each post LH-EEC time point from pre LH-EEC baseline score will be summarized. Individual data listings of all observed values will be presented by study group, visit and time points.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 or older in good general health on the basis of medical history and ophthalmic examination.
2. Confirmed absence of pregnancy according to a urine pregnancy test at screening (Visit 1) for WOCBP. WOCBP must agree to use effective methods of birth control during the study such as:

   * Oral, transdermal, injectable, vaginal ring, implantable contraceptives, intrauterine devices, or intrauterine system starting/placement at least 4 weeks prior to Screening (Visit 1)
   * Double barrier methods (diaphragm, cervical/vault cap, condom, contraceptive sponge plus a spermicide)
   * Having a sterile partner (vasectomized > 90 days prior to Screening Visit 1 )
   * Practicing abstinence
   * Non-heterosexual lifestyle
3. Subjects must have no known systemic disease or need for medication which may interfere with the study.
4. Subjects must have healthy eyes (no ophthalmic medication use nor current ocular infection) and concomitant medication may be permitted at the discretion of the investigator as long as there is no interference with study objectives or subject's safety.
5. Subjects must have VA best corrected to 20/50 or better for each eye (with Investigator discretion for subjects with amblyopia).
6. Subjects must be willing to discontinue their own contact lens wear for the period 7 days before Screening Visit 1 through to the end of the study.
7. Ability to comply with the study protocol, provide written consent and complete the study.

Exclusion Criteria:

1. Any ocular disease including keratoconus or nystagmus.
2. Any tarsal abnormalities or corneal neovascularization > Grade 2 (see Appendix 3).
3. Ocular surgery including refractive surgery within the last 12 months.
4. IOP >25 mmHg and utilization of any prescribed ophthalmic medication.
5. Subjects who fit the criteria for both ADDE and LDDE.
6. Clinically significant disease or abnormality which the Investigator may judge unsafe to participate in the study and/or interfere with the outcome of the study, including clinically significant physical findings on SLE or fundus evaluation.
7. Pregnancy or breastfeeding, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period, or for 30 days following the study period.
8. Subjects who require the use of antihistamines, corticosteroids or glaucoma medications on a regular basis and who are unwilling to discontinue the use of these medications for appropriate periods prior to the study visits.
9. Current participation in another clinical study involving an experimental product, or participation in such a study within 30 days prior to study entry.
10. Not meeting concomitant medication washouts.
11. Inability to discontinue any ophthalmic eye drops including over the counter (OTC) therapies.
12. Be an employee of the site that is directly involved in the management, administration, or support of this study or be an immediate family member of the same.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male and female volunteers, aged 18 years or older, either without or with DES (aqueous and lipid deficient).
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-03-11 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
To compare the clinical measurements of DES to the TFI measurements | Change from baseline to 120 minutes in the LH-EEC
  The correlation between the clinical measurements of DES and the corresponding TFI measurement of interest will evaluate the association between the two assessments.
To evaluate the repeatability of the TFI | Change from baseline after 30 minutes
  The repeatability of the TFI will be evaluated from summary of TFI assessments between Visit 2 and Visit 3. The sensitivity of the imager to detect changes in ocular surface integrity will be evaluated from the summary of baseline to post baseline assessment scores by time points and visit.
To evaluate the ability of the TFI to detect changes in ocular surface integrity during and after desiccation in a LH-EEC model. | Change from baseline measurements prior to entering the LH-EEC and at 15, 30, 60, 90, and 120 min (+5 min) after start of exposure to LH-EEC
  The sensitivity of the imager to detect changes in ocular surface integrity will be valuated from the summary of baseline to post baseline assessment scores by time points and visit.

SECONDARY OUTCOMES:
TFI lipid layer thickness (LLT) | Change from baseline measurements prior to entering the LH-EEC and at 15, 30, 60, 90, and 120 min (+5 min) after start of exposure to LH-EEC
  Lipid layer thickness in nanometers (nm) as measured by the Tear film Imager(TFI)
TFI aqueous layer thickness (ALT) | Change from baseline measurements prior to entering the LH-EEC and at 15, 30, 60, 90, and 120 min (+5 min) after start of exposure to LH-EEC
  Aqueous layer thickness in nanometers (nm) as measured by the Tear film Imager (TFI)
Schirmer's Test score | Change from baseline to 120 minutes in the LH-EEC
  Schirmer's Test score without anesthetic
Tear Break Up time (TBUT) | Change from baseline to 120 minutes in the LH-EEC
  Tear Break Up time (TBUT) with Fluorescein enhancement
TFI lipid break up time (LBUT) | Change from baseline measurements prior to entering the LH-EEC and at 15, 30, 60, 90, and 120 min (+5 min) after start of exposure to LH-EEC
  Lipid break up time (LBUT) as measured by the Tear Film Imager (TFI)
Total CFS | Change from baseline to 120 minutes in the LH-EEC
  Total score of Corneal Fluorescein Staining (CFS) over 2 regions
Total CLGS | Change from baseline to 120 minutes in the LH-EEC
  Total score of Conjunctival Lissamine Green Staining (CLGS) over 5 regions
Ocular Surface Disease Index (OSDI) | At baseline
  Total score of Ocular Surface Disease Index (OSDI) questionnaire
Dryness symptom score | Change from baseline measurements prior to entering the LH-EEC and at 15, 30, 60, 90, and 120 min (+15 min) after start of exposure to LH-EEC
  Collecting dryness symptom scores from subjects is a common clinical procedure in dry eye studies.
Total symptom score | Change from baseline measurements prior to entering the LH-EEC and at 15, 30, 60, 90, and 120 min (+15 min) after start of exposure to LH-EEC
  Collecting symptom scores from subjects is a common clinical procedure in dry eye studies.
Blink rate | Change from baseline measurements prior to entering the LH-EEC and at 15, 30, 60, 90, and 120 min (+15 min) after start of exposure to LH-EEC
  Blink rate will be assessed for both eyes together throughout the study.
Inter Blink Interval (IBI) | Change from baseline measurements prior to entering the LH-EEC and at 15, 30, 60, 90, and 120 min (+5 min) after start of exposure to LH-EEC
  Inter Blink Interval (IBI) as measured by the Tear Film Imager (TFI)
TFI field of view | Change from baseline measurements prior to entering the LH-EEC and at 15, 30, 60, 90, and 120 min (+5 min) after start of exposure to LH-EEC
  Field of view as measured by the Tear Film Imager (TFI)
TFI resolution | Change from baseline measurements prior to entering the LH-EEC and at 15, 30, 60, 90, and 120 min (+5 min) after start of exposure to LH-EEC
  Lipid lateral resolution as measured by the Tear Film Imager (TFI)

OTHER OUTCOMES:
Safety Analysis | At the study check out at the end of visit 3.
  Number of adverse events (AE) per group

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, MD, Principal Investigator — Inflamax Research Incorporated
Locations (1):
- Inflamax Research Inc., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No